CLINICAL TRIAL: NCT06631300
Title: A Randomized, Placebo-controlled Trial of Prednisone in Refractory Restless Legs Syndrome: a Pilot Study
Acronym: PrRLS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, J STEVEN POCETA, Principal Investigator, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-24-8351
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Restless Legs Syndrome
Keywords: refractory rls; rls; restless legs syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prednisone group (Experimental): A prednisone taper will be given to the subjects.
  Interventions: Drug: Prednisone
- Placebo group (Placebo Comparator): A placebo taper will be given to match the number of pills being tapered in the prednisone group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — A prednisone taper will be given to the subjects as follows: prednisone 40mg for 3 days, prednisone 30mg for 3 days, prednisone 20mg for 3 days, prednisone 10mg for 3 days, prednisone 5mg for 3 days, then off for a total of 15 days.
  Arms: Prednisone group
Drug: Placebo — A placebo taper will be given to match the same number of pills administered in each stage of the prednisone taper.
  Arms: Placebo group

SUMMARY:
Restless legs syndrome is a common sleep-related movement disorder that affects up to 15% of the population in North America, characterized by an uncomfortable urge to move the legs. This has been associated with poor quality of sleep and overall decreased quality of life. Chronic inflammation has been implicated as a key mediator of the low intracranial iron stores that characterize restless legs syndrome (RLS). Current medications for RLS target concomitant low serum iron levels or the dopaminergic pathway, but none target the inflammatory pathway. A novel therapy that focuses on inflammation would allow for additional research into the role of inflammation and cytokines in the development of RLS, and potentially unlock a new class of medications to treat patients with RLS. A small amount of prior evidence suggest that RLS symptoms improve with steroids, with associated improved quality of life, and with decreasing hepcidin levels as a biomarker of symptom severity. This pilot study, using an RCT design, serves to assess the efficacy of glucocorticoids in the alleviation of RLS symptoms, which would further anchor the association between RLS, inflammation, and one of its potential mediators - hepcidin. By giving a prednisone taper versus placebo, this study primarily aims to assess the effect of glucocorticoids on 1) decreasing RLS symptom severity. This study also aims to measure 2) objectively measured improvement in sleep, 3) changes in baseline and post-treatment hepcidin levels, and 4) prevalence of adverse events including psychosis and weight gain. RLS can be a debilitating disease and several non-traditional medications have been tested but with unequivocal results. Glucocorticoids may be an easily accessible and affordable key to better quality of life for RLS patients, especially those with refractory RLS.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Refractory RLS defined as restless legs unresponsive to monotherapy with tolerable doses of first-line agents due to reduction in efficacy, augmentation, or adverse effects
* IRLS score greater than 15

Exclusion Criteria:

* Pregnancy
* Prescence of iron deficiency anemia
* History of Diabetes Mellitus Type 1 and Type 2
* History of uncontrolled hypertension
* Presence of immunosuppression (HIV or currently taking immunosuppressants)
* Any prior adverse reaction to glucocorticoids
* History of dementia or major psychiatric diseases with psychosis
* Lack of ability to understand the experimental protocol and to adequately communicate in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group rating scale (IRLS) | Taken on Day 0, Day 14, and Day 21
  Evaluates severity of restless legs syndrome symptoms
Clinical Global Impression (CGI) | Taken on Day 0 and Day 21
  Participant quantifies overall severity of illness before and after intervention

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | Taken on Day 0 and Day 21
  Subjective measure of participant's sleepiness
Insomnia Severity Index (ISI) | Taken on Day 0 and Day 21
  Quantifies participant's perception of insomnia severity
Hepcidin levels | Taken on Day 0 and Day 21
  Measures serum hepcidin levels
Fitbit Sleep Score | Taken on Day 0 through Day 21
  Composite of sleep duration, sleep quality, and restoration as measured on Fitbit device based on heart rate variability
Generic Assessment of Side Effects (GASE) | Taken on Day 14, Day 21 and Day 35
  Monitors for study related complications

CONTACTS AND LOCATIONS:
Overall Officials: Mark Esguerra, MD, Study Chair — Scripps Health

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect patient privacy and confidentiality.